CLINICAL TRIAL: NCT02217293
Title: Efficacy of Pulsed Radiofrequency of the Median Nerve Under Ultrasound Guidance in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSGHIRB: 1-101-05-049
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Pulsed radiofrequency; Ultrasound-guided; Carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulsed Radiofrequency (Active Comparator): Pulsed radiofrequency (PRF) treatment, a relative novel pain intervention at recent decade, was found to be able to alleviate pain by delivering an electrical field and heat bursts at a temperature less than 42°C to neural tissue in the absence of neural injury
  Interventions: Device: Pulsed Radiofrequency
- Night splint (No Intervention): The wrist night splint was firmly fixed in a neutral position to immobilize the affected wrist. Patients were ordered to wear the splint while resting at night and at least 8 hours per day during the period of study

INTERVENTIONS:
Device: Pulsed Radiofrequency — Pulsed radiofrequency (PRF) treatment, a relative novel pain intervention at recent decade, was found to be able to alleviate pain by delivering an electrical field and heat bursts at a temperature less than 42°C to neural tissue in the absence of neural injury. The ultrasound-guided PRF was performed before night splint in intervention group.
  Other Names: Neurotherm NT1000, Neurotherm Inc., USA
  Arms: Pulsed Radiofrequency

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy. Although many conservative forms of management including the use of wrist splint, steroid injections and therapeutic ultrasound are applicable, their effectiveness is typically insignificant or short-lived.

Pulsed radiofrequency (PRF) treatment, a relative novel pain intervention at recent decade, was found to be able to alleviate pain for certain kinds of chronic pain conditions without damaging nerve. However, the application of PRF in CTS is scarce.

The purpose of this study was to assess the analgesic effect and prognosis of ultrasound-guided PRF in the median nerve in patients with CTS.

DETAILED DESCRIPTION:
Background and Purpose:

Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy. Although many conservative forms of management including the use of wrist splint, steroid injections and therapeutic ultrasound are applicable, their effectiveness is typically insignificant or short-lived.

Pulsed radiofrequency (PRF) treatment, a relative novel pain intervention at recent decade, was found to be able to alleviate pain for certain kinds of chronic pain conditions without damaging nerve. However, the application of PRF in CTS is scarce. The purpose of this study was to assess the analgesic effect and prognosis of ultrasound-guided PRF in the median nerve in patients with CTS.

Study design Duration: 2012/1/1 to 2012/12/31. Subjects: Outpatient subjects who had typical symptoms and signs of CTS, such as positive Tinel's sign or Phalen's test and numbness/tingling in at least two of the first, second, and third digits and were all confirmed by electrophysiological study, were considered and enrolled. The patients who had conditions mimicking CTS, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previous wrist surgery or steroid injection for CTS, were all excluded. Patient number: 40. Methods: The enrolled patients were randomized into two groups as the intervention group, who received one dose of PRF and the control group, who did not received RPF treatment by using drawing sealed envelope. To provide fundamental medical care of CTS, a wrist night splint was prescribed for each subject in both groups. Patients were ordered to wear the splint while resting at night and at least 8 hours per day during the period of study. All procedures were conducted by single physician. All the measurements were performed by single physician who was blinded for the randomization, and the evaluation time was performed before intervention as well as the 1st, 4th, 8th and 12th weeks after treatment. All patients were instructed to keep away from getting any other treatments for their pain or discomfort resulting from CTS including analgesic agents, injection or acupuncture etc. during the period of follow-up. They were asked to notify us if they had taken these therapies.

Outcome measurements:

1. Visual analog scale (VAS): The severity of digital pain during any activity most time per day was marked down in the pain scale. Each patient reported the VAS score every day at the same time after the initial treatment until 2 consecutive days reaching the definition of onset time which was defined as the day the VAS score had declined by 40% or more.
2. Boston Carpal Tunnel Syndrome Questionnaire (BCTQ).
3. Cross-sectional area of the median nerve: It was measured at the proximal inlet of the carpal tunnel (level with the pisiform bone) by the same physician.
4. Sensory nerve conduction velocity (SNCV) of median nerve.
5. Finger pinch. Data analysis: Demographic data were analyzed by the Mann-Whitney U test for continuous data and X2 test for categorical data. Wilcoxon's signed rank test was used to compare the outcome measures within each group of patients. The outcomes at each follow-up period were compared with the baseline values and differences between both groups were investigated using the Mann-Whitney U test. Comparability of change of VAS score and finger pinch measurements among the two groups was assessed using Mann-Whitney U test. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient subjects who had typical symptoms and signs of CTS, such as positive Tinel's sign or Phalen's test and numbness/tingling in at least two of the first, second, and third digits and were all confirmed by electrophysiological study, were considered and enrolled.

Exclusion Criteria:

* The patients who had conditions mimicking CTS, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previous wrist surgery or steroid injection for CTS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on1st, 4th, 8th and 12th weeks after treatment. | Pre-treatment, 1st, 4th, 8th and 12th weeks after treatment.
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 1st, 4th, 8th and 12th weeks after treatment. | Pre-treatment, 1st, 4th, 8th and 12th weeks after treatment.
  Using the Boston Carpal Tunnel Syndrome Questionnaire to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline in cross-sectional area of the median nerve on 1st, 4th, 8th and 12th weeks after treatment. | Pre-treatment, 1st, 4th, 8th and 12th weeks after treatment.
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline in conduction velocity, ampliture of median nerve on 1st, 4th, 8th and 12th weeks after treatment. | Pre-treatment, 1st, 4th, 8th and 12th weeks after treatment.
  The antidromic sensory nerve conduction velocityof the median nerve was performed on all subjects according to the protocol reported by the American Academy of Neurology with SierraWave, Cadwell (USA). The median nerve was stimulated at the wrist between the palmar longus and flexor carpal radialis tendon at a distance of approximately 14 cm from the active electrode.
Change from baseline in finger pinch on 1st, 4th, 8th and 12th weeks after treatment. | Pre-treatment, 1st, 4th, 8th and 12th weeks after treatment.
  The finger pinch strength was measured using Jamar dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Cheng Chen, MD, MS, Principal Investigator — Tri-Service General Hospital, School of Medicine, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, School of Medicine, National Defense Medical Center, Taipei, Neihu, Taiwan

REFERENCES:
- [Background] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. [Prevalence for clinically proved carpal tunnel syndrome is 4 percent]. Lakartidningen. 2000 Apr 5;97(14):1668-70. Swedish. PMID 10815392
- [Background] O'Connor D, Marshall S, Massy-Westropp N. Non-surgical treatment (other than steroid injection) for carpal tunnel syndrome. Cochrane Database Syst Rev. 2003;2003(1):CD003219. doi: 10.1002/14651858.CD003219. PMID 12535461
- [Background] Katz JN, Keller RB, Simmons BP, Rogers WD, Bessette L, Fossel AH, Mooney NA. Maine Carpal Tunnel Study: outcomes of operative and nonoperative therapy for carpal tunnel syndrome in a community-based cohort. J Hand Surg Am. 1998 Jul;23(4):697-710. doi: 10.1016/S0363-5023(98)80058-0. PMID 9708386
- [Background] Chua NH, Vissers KC, Sluijter ME. Pulsed radiofrequency treatment in interventional pain management: mechanisms and potential indications-a review. Acta Neurochir (Wien). 2011 Apr;153(4):763-71. doi: 10.1007/s00701-010-0881-5. Epub 2010 Nov 30. PMID 21116663
- [Result] Werner RA, Andary M. Carpal tunnel syndrome: pathophysiology and clinical neurophysiology. Clin Neurophysiol. 2002 Sep;113(9):1373-81. doi: 10.1016/s1388-2457(02)00169-4. PMID 12169318
- [Result] Haider N, Mekasha D, Chiravuri S, Wasserman R. Pulsed radiofrequency of the median nerve under ultrasound guidance. Pain Physician. 2007 Nov;10(6):765-70. PMID 17987099
- [Result] Wong SM, Griffith JF, Hui AC, Tang A, Wong KS. Discriminatory sonographic criteria for the diagnosis of carpal tunnel syndrome. Arthritis Rheum. 2002 Jul;46(7):1914-21. doi: 10.1002/art.10385. PMID 12124876
- [Derived] Chen LC, Ho CW, Sun CH, Lee JT, Li TY, Shih FM, Wu YT. Ultrasound-Guided Pulsed Radiofrequency for Carpal Tunnel Syndrome: A Single-Blinded Randomized Controlled Study. PLoS One. 2015 Jun 12;10(6):e0129918. doi: 10.1371/journal.pone.0129918. eCollection 2015. PMID 26067628